CLINICAL TRIAL: NCT02024828
Title: Feeding Readiness in Preterm Infants
Brief Title: Testing Four Feeding Approaches to Oral Feeding in Preterm Infants
Acronym: PRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01NR005182 (NIH)
Record Dates: First submitted 2013-12-19; First posted 2013-12-31 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2011-05

CONDITIONS: Preterm Infant
Keywords: Infant feeding
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Early/Slow (Experimental): Infants were offered oral feedings beginning at 32 weeks PMA. They were offered 2 oral feedings per day for 3 days (Days 1-3). The number of oral feedings offered per day increased by 1 feeding every other day until day 14 when they were offered 8 oral feedings each day (Days 4-5, 3 oral feeds offered; Days 6-7, 4 oral feeds offered; Days 8-9, 5 oral feeds offered; Days 10-11, 6 oral feeds offered; Days 12-13, 7 oral feeds offered; Day14, 8 oral feeds offered). Any feedings not offered orally were provided by gavage.
  Interventions: Other: Early/Slow
- Early/Fast (Experimental): Infants were first offered oral feedings beginning at 32 weeks PMA. They were offered 8 oral feedings every day, at each of 8 scheduled daily feedings.
  Interventions: Other: Early/Fast
- Late/Slow (Experimental): Infants were offered oral feedings beginning at 34 weeks PMA. They were offered 2 oral feedings per day for 3 days (Days 1-3). The number of oral feedings offered per day increased by 1 feeding every other day until day 14 when they were offered 8 oral feedings each day (Days 4-5, 3 oral feeds offered; Days 6-7, 4 oral feeds offered; Days 8-9, 5 oral feeds offered; Days 10-11, 6 oral feeds offered; Days 12-13, 7 oral feeds offered; Day14, 8 oral feeds offered). Any feedings not offered orally were provided by gavage.
  Interventions: Other: Late/Slow
- Late/Fast (Experimental): Infants were offered oral feedings beginning at 34 weeks PMA. They were offered 8 oral feedings every day, at each of 8 scheduled daily feedings.
  Interventions: Other: Late/Fast

INTERVENTIONS:
Other: Early/Slow
  Arms: Early/Slow
Other: Early/Fast
  Arms: Early/Fast
Other: Late/Slow
  Arms: Late/Slow
Other: Late/Fast
  Arms: Late/Fast

SUMMARY:
The purpose of this study was to test the effect of four randomly assigned approaches to oral feeding transition on feeding outcomes in preterm infants.

DETAILED DESCRIPTION:
The study is completed.

ELIGIBILITY:
Inclusion Criteria:

* 1) the infant's gestational age at birth was less than 32 weeks; 2) the infant was receiving enteral feedings every three hours; 3) the infant was able medically to feed orally by 32 weeks post-menstrual age (PMA); and 3) the parents gave consent for the infant's participation.

Exclusion Criteria:

* 1) they were unable to begin oral feeding at 32 weeks PMA due to gastrointestinal, craniofacial, cardiovascular, neuromuscular, and/or genetic defects; 2) had surgical necrotizing enterocolitis; or 3) needed ventilator support, including nasal continuous positive airway pressure (CPAP), beyond 32 weeks PMA. Infants receiving oxygen by cannula were included.

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 109 (Actual)
Dates: Start 2006-07; Primary Completion 2011-01 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Feeding Performance | One oral feeding a day for 14 days
  Includes 3 components: Proportion consumed (volume taken/volume ordered), rate of consumption (volume consumed/minutes of feeding); proficiency (volume taken in first 5 minutes of feeding/volume ordered)

SECONDARY OUTCOMES:
Clinical outcomes | Participants will be followed for the duration of the hospital stay, an expected average from starting oral feedings of 3 weeks
  Days to discharge from first oral feeding
Post-discharge feeding | 2 weeks after discharge
  Performance at feeding 2 weeks after hospital discharge using the Early Infant Feeding Scale, an observational tool of infant feeding behaviors

CONTACTS AND LOCATIONS:
Locations (1):
- CCHMC, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Alberts JR, Pickler RH. Evolution and development of dual ingestion systems in mammals: notes on a new thesis and its clinical implications. Int J Pediatr. 2012;2012:730673. doi: 10.1155/2012/730673. Epub 2012 Sep 18. PMID 23028391
- [Background] Pickler RH, McGrath JM, Reyna BA, McCain N, Lewis M, Cone S, Wetzel P, Best A. A model of neurodevelopmental risk and protection for preterm infants. J Perinat Neonatal Nurs. 2010 Oct-Dec;24(4):356-65. doi: 10.1097/JPN.0b013e3181fb1e70. PMID 21045616
- [Result] Pickler RH, Reyna BA, Griffin JB, Lewis M, Thompson AM. Changes in Oral Feeding in Preterm Infants Two Weeks After Hospital Discharge. Newborn Infant Nurs Rev. 2012 Dec 1;12(4):202-206. doi: 10.1053/j.nainr.2012.09.012. Epub 2012 Nov 15. PMID 23185127
- [Result] Pickler RH, McGrath JM, Reyna BA, Tubbs-Cooley HL, Best AM, Lewis M, Cone S, Wetzel PA. Effects of the neonatal intensive care unit environment on preterm infant oral feeding. Res Rep Neonatol. 2013 Apr 3;2013(3):15-20. doi: 10.2147/RRN.S41280. PMID 25552910